CLINICAL TRIAL: NCT07010172
Title: Effectiveness of Cognitive Rehabilitation Software in Female Patients With Fibromyalgia
Brief Title: Fibromyalgia, Cognitive Rehabilitation Software
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Savaş Karpuz (Other Government)
Responsible Party: Sponsor-Investigator, Savaş Karpuz, Associate Professor, Konya Beyhekim Training and Research Hospital
Organization: Konya Beyhekim Training and Research Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-79735520-799
Record Dates: First submitted 2025-05-02; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia; Cognitive Rehabilitation
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cognitive rehabilitation software (Experimental): 3-5 sessions per week, 4 weeks cognitive rehabilitation with computer software
  Interventions: Device: cognitive rehabilitation with computer software

INTERVENTIONS:
Device: cognitive rehabilitation with computer software — 3-5 sessions per week, 4 weeks cognitive rehabilitation with computer software

SUMMARY:
In recent years, especially in developed countries, FMS has emerged as a serious social problem by decreasing labour force and quality of life. Especially clinicians have started to consider cognitive dysfunction in FMS as a separate clinical condition. In the light of the data obtained, can say that cognitive dysfunction increases in the presence of depression, anxiety, sleep disorders, endocrine imbalances and pain.

Neuroscience and technological advances make it possible to meet the demand for care and improve the quality of stimulation by enabling the automation of many cognitive training procedures, improving patient record reliability and optimising performance of disability functions. The recently implemented RehaCom and HeadApp programmes (Schuhfried, Austria). excellent results have been reported in clinical practice with no significant adverse effects.

This study will investigate the effectiveness of a cognitive rehabilitation programme using computer software in female patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Diagnosed with fibromyalgia
* 18-65 years old

Exclusion Criteria:

* concomitant neurological disorder, learning disorder or cognitive impairment
* current alcohol or recreational drug dependence or long-term (≥5 years) history of substance abuse
* visual or hearing impairment that would interfere with cognitive testing
* diagnosis of untreated obstructive sleep apnoea,
* atypical sleep/wake patterns (e.g. night shift workers)
* Lack of computer and internet access

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Stroop Colour and Word Test | start and first month
Number Range Test | start and first month

SECONDARY OUTCOMES:
modified Fibromyalgia impact questionnaire | start and first month

IPD SHARING:
Plan to Share IPD: No